CLINICAL TRIAL: NCT05751499
Title: Diagnostic and Prognostic Blood Markers in Non Specific Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Collaborators: KRL Hospital, Islamabad (Other)
Responsible Party: Sponsor
Other Study IDs: Rana Muhammad Tahir
Record Dates: First submitted 2022-12-17; First posted 2023-03-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CASE GROUP: 1. Both male & Female patients
  2. Age group 18-60 Years
  3. Diagnosed with nonspecific low back pain in acute/flared stage
  Interventions: Diagnostic Test: • Blood Markers CRP, TNFα, IL-6, IL-8, IL-1, and IL-1β AND FIBRINOGEN
- CONTROL GROUP: MALE AND FEMALE AGE GROUP 18 TO 60 YEARS NOT SUFFERING FROM LOW BACK PAIN
  Interventions: Diagnostic Test: • Blood Markers CRP, TNFα, IL-6, IL-8, IL-1, and IL-1β AND FIBRINOGEN

INTERVENTIONS:
Diagnostic Test: • Blood Markers CRP, TNFα, IL-6, IL-8, IL-1, and IL-1β AND FIBRINOGEN — * Low Back Outcome Scale
  * Center for Epidemiological Studies-Depression Scale (CES-D)
  * International Physical Activity Questionnaire
  * Roland-Morris Disability Questionnaire
  * Force Platform
  * Pain Self-Efficacy Questionnaire (PSEQ)
  * Numeric Rating Scale
  * Job Content Questionnaire
  * Pits Burgh Sleep Quality Index (PSQI)
  * Orebo Musculoskeletal Pain Screening Questionnaire
  * Gait & Balance App
  * Keele STarT Back Screening Tool (SBST)
  * Fear-Avoidance Beliefs Questionnaire (FABQ)
  * Pain Catastrophizing Scale

SUMMARY:
• To compare the diagnostic and prognostic blood markers in acute and chronic nonspecific low back pain with healthy controls

DETAILED DESCRIPTION:
* To compare the diagnostic and prognostic blood markers in acute and chronic nonspecific low back pain with healthy controls
* To predict the diagnostic and prognostic blood markers on sleep, depression and anxiety in acute and chronic non specific low back pain.
* To compare the effect of physical activity with blood markers in acute and chronic non specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Both male & Female patients
2. Age group 18-60 Years
3. Diagnosed with nonspecific low back pain in acute/flared stage

Exclusion Criteria:

* Any serious conditions like neurological conditions
* Any infection
* Tumor
* Spinal Surgery
* Cognitive Impairments
* Refusal to sign consent
* patients taking any type of psychological management or rheumatologic disease would be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: PEOPLE BETWEEN 18 TO 60 YEARS HAVING LOW BACK PAIN WITH NON SPECIFIC REASON
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
CRP | 0 weeks [at the start of data]
  It measures the level of C-reactive proteins in a sample of blood. CRP is a protein made by lever. It shows inflammation in the body
CRP | 8th weeks
  It measures the level of C-reactive proteins in a sample of blood. CRP is a protein made by lever. It shows inflammation in the body
CRP | 16th weeks
  It measures the level of C-reactive proteins in a sample of blood. CRP is a protein made by lever. It shows inflammation in the body
CRP | 24th weeks
  It measures the level of C-reactive proteins in a sample of blood. CRP is a protein made by lever. It shows inflammation in the body
TNF ALPHA | 0 weeks
  TNF ALPHA is an adipokine and a cytokine. It is one of the most important pro-inflammatory cytokine.
TNF ALPHA | 8 weeks
  TNF ALPHA is an adipokine and a cytokine. It is one of the most important pro-inflammatory cytokine.
TNF ALPHA | 16 weeks
  TNF ALPHA is an adipokine and a cytokine. It is one of the most important pro-inflammatory cytokine.
TNF ALPHA | 24 weeks
  TNF ALPHA is an adipokine and a cytokine. It is one of the most important pro-inflammatory cytokine.
IL 1 | 0 weeks
  Interleukin-1 is a group of 11 cytokines that plays a central role in the regulation of immune and inflammatory response to infections
IL 1 | 8 weeks
  Interleukin-1 is a group of 11 cytokines that plays a central role in the regulation of immune and inflammatory response to infections
IL 1 | 16 weeks
  Interleukin-1 is a group of 11 cytokines that plays a central role in the regulation of immune and inflammatory response to infections
IL 1 | 24 weeks
  Interleukin-1 is a group of 11 cytokines that plays a central role in the regulation of immune and inflammatory response to infections
IL 6 | 0 weeks
  Interleukin-6 promptly and transiently produced in response to infections and tissues injuries.
IL 6 | 8 weeks
  Interleukin-6 promptly and transiently produced in response to infections and tissues injuries.
IL 6 | 16 weeks
  Interleukin-6 promptly and transiently produced in response to infections and tissues injuries.
IL 6 | 24 weeks
  Interleukin-6 promptly and transiently produced in response to infections and tissues injuries.
IL-8 | 0 weeks
  Interleukin-8 is a chemoattractant cytokine produced by variety of tissues and blood cells. It activates neutrophils in inflammatory regions
IL-8 | 8 weeks
  Interleukin-8 is a chemoattractant cytokine produced by variety of tissues and blood cells. It activates neutrophils in inflammatory regions
IL-8 | 16 weeks
  Interleukin-8 is a chemoattractant cytokine produced by variety of tissues and blood cells. It activates neutrophils in inflammatory regions
IL-8 | 24 weeks
  Interleukin-8 is a chemoattractant cytokine produced by variety of tissues and blood cells. It activates neutrophils in inflammatory regions
IL-1 BETA | 0 weeks
  IL-1Beta is a pro inflammatory cytokine implicated in pain, inflammation and autoimmune condition
IL-1 BETA | 8 weeks
  IL-1Beta is a pro inflammatory cytokine implicated in pain, inflammation and autoimmune condition
IL-1 BETA | 16 weeks
  IL-1Beta is a pro inflammatory cytokine implicated in pain, inflammation and autoimmune condition
IL-1 BETA | 24 weeks
  IL-1Beta is a pro inflammatory cytokine implicated in pain, inflammation and autoimmune condition
Fibrinogen | 0 weeks
  Fibrinogen is a protein produced by liver, its high levels may occur as a part of normal response to infection or inflammation.
Fibrinogen | 8 weeks
  Fibrinogen is a protein produced by liver, its high levels may occur as a part of normal response to infection or inflammation.
Fibrinogen | 16 weeks
  Fibrinogen is a protein produced by liver, its high levels may occur as a part of normal response to infection or inflammation.
Fibrinogen | 24 weeks
  Fibrinogen is a protein produced by liver, its high levels may occur as a part of normal response to infection or inflammation.

SECONDARY OUTCOMES:
Numeric rating scale | 0 weeks
  Self-reported pain intensity will be measured using an 11-point NRS ranging from "none" to "worst imaginable pain
Numeric rating scale | 8 weeks
  Self-reported pain intensity will be measured using an 11-point NRS ranging from "none" to "worst imaginable pain
Numeric rating scale | 16 weeks
  Self-reported pain intensity will be measured using an 11-point NRS ranging from "none" to "worst imaginable pain
Numeric rating scale | 24 weeks
  Self-reported pain intensity will be measured using an 11-point NRS ranging from "none" to "worst imaginable pain
Low Back outcome scale | 0 weeks
  The Low Back outcome scale evaluates pain and physical function. It has a score in the range from 0 to 75 and the higher score indicates better condition. It categorizes patients into a 4-grade classification scheme: excellent ≥65; good 50-64; fair 30-49, and poor 0-29.
Low Back outcome scale | 8 weeks
  The Low Back outcome scale evaluates pain and physical function. It has a score in the range from 0 to 75 and the higher score indicates better condition. It categorizes patients into a 4-grade classification scheme: excellent ≥65; good 50-64; fair 30-49, and poor 0-29.
Low Back outcome scale | 16 weeks
  The Low Back outcome scale evaluates pain and physical function. It has a score in the range from 0 to 75 and the higher score indicates better condition. It categorizes patients into a 4-grade classification scheme: excellent ≥65; good 50-64; fair 30-49, and poor 0-29.
Low Back outcome scale | 24 weeks
  The Low Back outcome scale evaluates pain and physical function. It has a score in the range from 0 to 75 and the higher score indicates better condition. It categorizes patients into a 4-grade classification scheme: excellent ≥65; good 50-64; fair 30-49, and poor 0-29.
Center for Epidemiological Studies-Depression Scale (CES-D): | 0 weeks
  Centre for epidemiological studies of depression scale (CES-D) evaluates depressive symptoms. It has score range of 0 to 60 with higher score indicating increased depressive symptoms.
Center for Epidemiological Studies-Depression Scale (CES-D): | 8 weeks
  Centre for epidemiological studies of depression scale (CES-D) evaluates depressive symptoms. It has score range of 0 to 60 with higher score indicating increased depressive symptoms.
Center for Epidemiological Studies-Depression Scale (CES-D): | 16 weeks
  Centre for epidemiological studies of depression scale (CES-D) evaluates depressive symptoms. It has score range of 0 to 60 with higher score indicating increased depressive symptoms.
Center for Epidemiological Studies-Depression Scale (CES-D): | 24 weeks
  Centre for epidemiological studies of depression scale (CES-D) evaluates depressive symptoms. It has score range of 0 to 60 with higher score indicating increased depressive symptoms.
Pain catastrophizing scale | 0 weeks
  Pain catastrophizing scale is used for measuring catastrophic thinking related to pain. The total score ranges from 0-52, along with three subscale scores assessing rumination, magnification and helplessness
Pain catastrophizing scale | 8 weeks
  Pain catastrophizing scale is used for measuring catastrophic thinking related to pain. The total score ranges from 0-52, along with three subscale scores assessing rumination, magnification and helplessness
Pain catastrophizing scale | 16 weeks
  Pain catastrophizing scale is used for measuring catastrophic thinking related to pain. The total score ranges from 0-52, along with three subscale scores assessing rumination, magnification and helplessness
Pain catastrophizing scale | 24 weeks
  Pain catastrophizing scale is used for measuring catastrophic thinking related to pain. The total score ranges from 0-52, along with three subscale scores assessing rumination, magnification and helplessness
Fear-Avoidance Beliefs Questionnaire (FABQ) | 0 weeks
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which measures patients' fear of pain and consequent avoidance of physical activity because of their fear. It is a 7-point Likert scale where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Fear-Avoidance Beliefs Questionnaire (FABQ) | 8 weeks
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which measures patients' fear of pain and consequent avoidance of physical activity because of their fear. It is a 7-point Likert scale where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Fear-Avoidance Beliefs Questionnaire (FABQ) | 16 weeks
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which measures patients' fear of pain and consequent avoidance of physical activity because of their fear. It is a 7-point Likert scale where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Fear-Avoidance Beliefs Questionnaire (FABQ) | 24 weeks
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which measures patients' fear of pain and consequent avoidance of physical activity because of their fear. It is a 7-point Likert scale where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Pain Self-Efficacy Questionnaire (PSEQ) | 0 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain.
Pain Self-Efficacy Questionnaire (PSEQ) | 8 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain.
Pain Self-Efficacy Questionnaire (PSEQ) | 16 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain.
Pain Self-Efficacy Questionnaire (PSEQ) | 24 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain.
Job Content Questionnaire | 0 weeks
  It is a questionnaire-based instrument designed to measure the "content" of a respondent's work tasks in a general manner which is applicable to all jobs and jobholders. It consists of 27 items quantified on a four-point Likert scale ranging from 1 (totally disagree) to 4 (totally agree).
Job Content Questionnaire | 8 weeks
  It is a questionnaire-based instrument designed to measure the "content" of a respondent's work tasks in a general manner which is applicable to all jobs and jobholders. It consists of 27 items quantified on a four-point Likert scale ranging from 1 (totally disagree) to 4 (totally agree).
Job Content Questionnaire | 16 weeks
  It is a questionnaire-based instrument designed to measure the "content" of a respondent's work tasks in a general manner which is applicable to all jobs and jobholders. It consists of 27 items quantified on a four-point Likert scale ranging from 1 (totally disagree) to 4 (totally agree).
Job Content Questionnaire | 24 weeks
  It is a questionnaire-based instrument designed to measure the "content" of a respondent's work tasks in a general manner which is applicable to all jobs and jobholders. It consists of 27 items quantified on a four-point Likert scale ranging from 1 (totally disagree) to 4 (totally agree).
Pittsburgh Sleep Quality Index (PSQI) | 0 week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. It has a score range of 0-21 where higher score indicates poor sleep.
Pittsburgh Sleep Quality Index (PSQI) | 8 week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. It has a score range of 0-21 where higher score indicates poor sleep.
Pittsburgh Sleep Quality Index (PSQI) | 16 week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. It has a score range of 0-21 where higher score indicates poor sleep.
Pittsburgh Sleep Quality Index (PSQI) | 24 week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. It has a score range of 0-21 where higher score indicates poor sleep.
International Physical Activity Questionnaire | 0 weeks
  IPAQ evaluates the health-related physical activity. Higher score indicates increased physical activity.
International Physical Activity Questionnaire | 8 weeks
  IPAQ evaluates the health-related physical activity. Higher score indicates increased physical activity.
International Physical Activity Questionnaire | 16 weeks
  IPAQ evaluates the health-related physical activity. Higher score indicates increased physical activity.
International Physical Activity Questionnaire | 24 weeks
  IPAQ evaluates the health-related physical activity. Higher score indicates increased physical activity.
Roland-Morris Disability Questionnaire | 0 weeks
  Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain.(18) The score ranges from 0 (no disability) to 11, 18 or 24 (max. disability) depending on the questionnaire that is used.
Roland-Morris Disability Questionnaire | 8 weeks
  Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain.(18) The score ranges from 0 (no disability) to 11, 18 or 24 (max. disability) depending on the questionnaire that is used.
Roland-Morris Disability Questionnaire | 16 weeks
  Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain.(18) The score ranges from 0 (no disability) to 11, 18 or 24 (max. disability) depending on the questionnaire that is used.
Roland-Morris Disability Questionnaire | 24 weeks
  Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain.(18) The score ranges from 0 (no disability) to 11, 18 or 24 (max. disability) depending on the questionnaire that is used.
Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ) | 0 weeks
  The ÖMPQ is a screening questionnaire used to predict long term disability and failure to return to work due to personal and environmental factors. The ÖMPQ score is used as a predictor of risk of long-term disability and failed return to work, with a higher score indicating higher risk.
Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ) | 8 weeks
  The ÖMPQ is a screening questionnaire used to predict long term disability and failure to return to work due to personal and environmental factors. The ÖMPQ score is used as a predictor of risk of long-term disability and failed return to work, with a higher score indicating higher risk.
Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ) | 16 weeks
  The ÖMPQ is a screening questionnaire used to predict long term disability and failure to return to work due to personal and environmental factors. The ÖMPQ score is used as a predictor of risk of long-term disability and failed return to work, with a higher score indicating higher risk.
Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ) | 24 weeks
  The ÖMPQ is a screening questionnaire used to predict long term disability and failure to return to work due to personal and environmental factors. The ÖMPQ score is used as a predictor of risk of long-term disability and failed return to work, with a higher score indicating higher risk.
Keele STarT Back Screening Tool (SBST) | 0 weeks
  The Keele STarT Back Screening Tool (SBST) (9-item version) is a brief validated tool, designed to screen primary care patients with low back pain for prognostic indicators that are relevant to initial decision making. It helps primary care clinicians to group patients into three categories of risk of poor outcome - low, medium, and high-risk.
Keele STarT Back Screening Tool (SBST) | 8 weeks
  The Keele STarT Back Screening Tool (SBST) (9-item version) is a brief validated tool, designed to screen primary care patients with low back pain for prognostic indicators that are relevant to initial decision making. It helps primary care clinicians to group patients into three categories of risk of poor outcome - low, medium, and high-risk.
Keele STarT Back Screening Tool (SBST) | 16 weeks
  The Keele STarT Back Screening Tool (SBST) (9-item version) is a brief validated tool, designed to screen primary care patients with low back pain for prognostic indicators that are relevant to initial decision making. It helps primary care clinicians to group patients into three categories of risk of poor outcome - low, medium, and high-risk.
Keele STarT Back Screening Tool (SBST) | 24 weeks
  The Keele STarT Back Screening Tool (SBST) (9-item version) is a brief validated tool, designed to screen primary care patients with low back pain for prognostic indicators that are relevant to initial decision making. It helps primary care clinicians to group patients into three categories of risk of poor outcome - low, medium, and high-risk.
Tampa Scale of Kinesiophobia (TSK) | 0 weeks
  It is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale ranges from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Tampa Scale of Kinesiophobia (TSK) | 8 weeks
  It is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale ranges from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Tampa Scale of Kinesiophobia (TSK) | 16 weeks
  It is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale ranges from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Tampa Scale of Kinesiophobia (TSK) | 24 weeks
  It is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale ranges from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Coping Strategies Questionnaire | 0 weeks
  The Coping Strategies Questionnaire (CSQ) is a 27-item tool which was developed in 1983 and it reflect the coping strategies frequently reported by patients in the management of pain.
Coping Strategies Questionnaire | 8 weeks
  The Coping Strategies Questionnaire (CSQ) is a 27-item tool which was developed in 1983 and it reflect the coping strategies frequently reported by patients in the management of pain.
Coping Strategies Questionnaire | 16 weeks
  The Coping Strategies Questionnaire (CSQ) is a 27-item tool which was developed in 1983 and it reflect the coping strategies frequently reported by patients in the management of pain.
Coping Strategies Questionnaire | 24 weeks
  The Coping Strategies Questionnaire (CSQ) is a 27-item tool which was developed in 1983 and it reflect the coping strategies frequently reported by patients in the management of pain.
Chronic Pain Grade Scale | 0 weeks
  The CPGS is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. It has 7 items. Subscale scores for pain intensity and disability are combined to calculate a chronic pain grade that enables classification of chronic pain patients into 5 hierarchical categories: grades 0 (no pain) to IV (high disability-severely limiting): grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting
Chronic Pain Grade Scale | 8 weeks
  The CPGS is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. It has 7 items. Subscale scores for pain intensity and disability are combined to calculate a chronic pain grade that enables classification of chronic pain patients into 5 hierarchical categories: grades 0 (no pain) to IV (high disability-severely limiting): grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting
Chronic Pain Grade Scale | 16 weeks
  The CPGS is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. It has 7 items. Subscale scores for pain intensity and disability are combined to calculate a chronic pain grade that enables classification of chronic pain patients into 5 hierarchical categories: grades 0 (no pain) to IV (high disability-severely limiting): grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting
Chronic Pain Grade Scale | 24 weeks
  The CPGS is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. It has 7 items. Subscale scores for pain intensity and disability are combined to calculate a chronic pain grade that enables classification of chronic pain patients into 5 hierarchical categories: grades 0 (no pain) to IV (high disability-severely limiting): grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting
Hospital Anxiety and Depression Scale | 0 weeks
  It is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients and measure symptoms of anxiety and depression. The questionnaire comprises seven questions for anxiety and seven questions for depression, and score ranges from 8 (mild) to 21 (severe symptoms).
Hospital Anxiety and Depression Scale | 8 weeks
  It is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients and measure symptoms of anxiety and depression. The questionnaire comprises seven questions for anxiety and seven questions for depression, and score ranges from 8 (mild) to 21 (severe symptoms).
Hospital Anxiety and Depression Scale | 16 weeks
  It is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients and measure symptoms of anxiety and depression. The questionnaire comprises seven questions for anxiety and seven questions for depression, and score ranges from 8 (mild) to 21 (severe symptoms).
Hospital Anxiety and Depression Scale | 24 weeks
  It is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients and measure symptoms of anxiety and depression. The questionnaire comprises seven questions for anxiety and seven questions for depression, and score ranges from 8 (mild) to 21 (severe symptoms).

OTHER OUTCOMES:
Gait & Balance App: | 0 weeks
  Using the Iphone 6 plus, this app will be installed in the phone and it will be used to measure balance and gait parameters. The phone will be fixed to patient's back with a securing balance during the performance of tasks
Gait & Balance App: | 8 weeks
  Using the Iphone 6 plus, this app will be installed in the phone and it will be used to measure balance and gait parameters. The phone will be fixed to patient's back with a securing balance during the performance of tasks
Gait & Balance App: | 16 weeks
  Using the Iphone 6 plus, this app will be installed in the phone and it will be used to measure balance and gait parameters. The phone will be fixed to patient's back with a securing balance during the performance of tasks
Gait & Balance App: | 24 weeks
  Using the Iphone 6 plus, this app will be installed in the phone and it will be used to measure balance and gait parameters. The phone will be fixed to patient's back with a securing balance during the performance of tasks
Force Platform | 0 weeks
  Force platform (Pasco PASPORT force platform-PS2141) will be used to analyze the patient's data for standing postural control. This platform has shown good reliability and validity. It will be measured with participants standing barefoot and blindfolded on a force plate for 75s. To test the effect of disruption of proprioception at the calf and lower back, the task will be repeated with vibrators (~ 60 Hz, 1 mm amplitude) attached bilaterally over the Achilles tendon and lumbar paraspinal muscles, separately, in random order. Vibrators will be switched on for 15 s at ~ 15 s after the start of the trial. Coordinates of CoP will be recorded
Force Platform | 8 weeks
  Force platform (Pasco PASPORT force platform-PS2141) will be used to analyze the patient's data for standing postural control. This platform has shown good reliability and validity. It will be measured with participants standing barefoot and blindfolded on a force plate for 75s. To test the effect of disruption of proprioception at the calf and lower back, the task will be repeated with vibrators (~ 60 Hz, 1 mm amplitude) attached bilaterally over the Achilles tendon and lumbar paraspinal muscles, separately, in random order. Vibrators will be switched on for 15 s at ~ 15 s after the start of the trial. Coordinates of CoP will be recorded
Force Platform | 16 weeks
  Force platform (Pasco PASPORT force platform-PS2141) will be used to analyze the patient's data for standing postural control. This platform has shown good reliability and validity. It will be measured with participants standing barefoot and blindfolded on a force plate for 75s. To test the effect of disruption of proprioception at the calf and lower back, the task will be repeated with vibrators (~ 60 Hz, 1 mm amplitude) attached bilaterally over the Achilles tendon and lumbar paraspinal muscles, separately, in random order. Vibrators will be switched on for 15 s at ~ 15 s after the start of the trial. Coordinates of CoP will be recorded
Force Platform | 24 weeks
  Force platform (Pasco PASPORT force platform-PS2141) will be used to analyze the patient's data for standing postural control. This platform has shown good reliability and validity. It will be measured with participants standing barefoot and blindfolded on a force plate for 75s. To test the effect of disruption of proprioception at the calf and lower back, the task will be repeated with vibrators (~ 60 Hz, 1 mm amplitude) attached bilaterally over the Achilles tendon and lumbar paraspinal muscles, separately, in random order. Vibrators will be switched on for 15 s at ~ 15 s after the start of the trial. Coordinates of CoP will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Waqar A Awan, PhD, Study Director — Faculty of Rehabilitation & Allied Health Sciences, Riphah International University; IMRAN AMJAD, PhD, Principal Investigator — Riphah International University
Locations (1):
- KRL Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No